CLINICAL TRIAL: NCT01282138
Title: A Study to Assess Alcon's Ocular Image Quantification Using Conjunctival Allergan Provocation Testing (CAPT) and Natural Allergen Exposure in an Environmental Exposure Chamber (EEC)
Brief Title: Assessment of Alcon's Ocular Image Quantification System
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: RDG-10-278
Record Dates: First submitted 2011-01-20; First posted 2011-01-24 (Estimated); Results first posted 2012-07-25 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-07

CONDITIONS: Allergic Conjunctivitis
Keywords: Allergic conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Olopatadine Hydrochloride; Ophthalmic Solutions; Dextrans; Hypromellose Derivatives; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patanol (Experimental): One drop twice daily in each eye for five days prior to allergen provocation testing, followed by an additional drop in each eye approximately 15 minutes prior to start of testing.
  Interventions: Drug: Olopatadine hydrochloride, 0.1% ophthalmic solution (Patanol)
- Tears Naturale II (Placebo Comparator): One drop twice daily in each eye for five days prior to allergen provocation testing, followed by an additional drop in each eye approximately 15 minutes prior to start of testing.
  Interventions: Other: Dextran 70 0.1%, hydroxypropyl methylcellulose 0.3% (Tears Naturale II)

INTERVENTIONS:
Drug: Olopatadine hydrochloride, 0.1% ophthalmic solution (Patanol) — One drop twice daily in each eye for 5 days, followed by an additional drop in each eye prior to allergen test.
  Other Names: Patanol®
  Arms: Patanol
Other: Dextran 70 0.1%, hydroxypropyl methylcellulose 0.3% (Tears Naturale II) — One drop twice daily in each eye for 5 days, followed by an additional drop in each eye prior to allergen test.
  Other Names: Tears Naturale II
  Arms: Tears Naturale II

SUMMARY:
The purpose of this study was to evaluate ocular responses with different allergen provocation methods.

DETAILED DESCRIPTION:
Subjects demonstrating a successful allergen response to a common allergen received the first study treatment and used as instructed for 5 days, after which they entered the Environmental Exposure Chamber (EEC) for a 3-hour exposure to a known concentration of the allergen. After waiting at least 7 days, subjects received the second study treatment and used as instructed for 5 days, after which a 3-hour Conjunctival Allergen Provocation Test (CAPT) was performed with an escalating concentration of the allergen. Subjects dosed with study treatment approximately 15 minutes prior to each allergen provocation test.

ELIGIBILITY:
Inclusion Criteria:

* History of allergic conjunctivitis;
* Active signs and symptoms of ocular allergies;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* History of dry eye;
* Presence of ocular infection;
* Presence of severe or serious ocular conditions;
* Symptoms of allergic conjunctivitis;
* Use of topical or systemic ocular medications as specified in protocol;
* Ocular surgery or laser surgery within 6 months of study start;
* Unwilling to discontinue contact lens wear 72 hours prior to Visit 1 and during study period;
* Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from one study center in Canada.
Period: EEC
Arm/Group | Patanol | Tears Naturale II
Started | 6 | 7
Completed | 6 | 7
Not Completed | 0 | 0
Period: CAPT
Arm/Group | Patanol | Tears Naturale II
Started | 6 | 7
Completed | 6 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patanol | Tears Naturale II | Total
Number analyzed (Participants) | 6 | 7 | 13
Age Continuous [Mean (Standard Deviation); unit: years] | 36.0 (10.4) | 39.9 (11.2) | 38.1 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  Canada | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Patient-Assessed Ocular Itching, Environmental Exposure Chamber (EEC), at 3 Hours
Description: As assessed by the participant after 3 hours in the EEC. Ocular itching was graded on a 0-4 scale, where 0=none, 1=tickling sensation involving one or more corners of the eye, 2=all over tickling sensation; 3=moderate continuous itching with desire to rub; 4=severe itching with irresistible urge to rub.
Time Frame: Baseline, 3 hours
Population: All enrolled participants
Measure: Mean (Standard Error); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | Patanol | Tears Naturale II
Number analyzed (Participants) | 6 | 7
Number analyzed (eyes) | 12 | 14
Units on a scale | -1.63 (0.6) | -1.11 (0.2)

2. Primary Outcome: Change From Baseline in Patient-Assessed Ocular Itching, Conjunctival Allergen Provocation Test (CAPT), at 3 Hours
Description: As assessed by the participant after 3 hours of CAPT. Ocular itching was graded on a 0-4 scale, where 0=none, 1=tickling sensation involving one or more corners of the eye, 2=all over tickling sensation; 3=moderate continuous itching with desire to rub; 4=severe itching with irresistible urge to rub.
Time Frame: Baseline, 3 hours
Population: All enrolled participants
Measure: Mean (Standard Error); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | Patanol | Tears Naturale II
Number analyzed (Participants) | 6 | 7
Number analyzed (eyes) | 12 | 14
Units on a scale | -0.38 (0.6) | -1.15 (0.5)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study: 3 months, 1 week, 6 days.
Description: This reporting group includes all enrolled subjects.
Arm/Group | Patanol | Tears Naturale II
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 0/6 | 2/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patanol (N=6) | Tears Naturale II (N=7)
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 — Not related
Intermittent Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Not related
Hordeolum Right Eye (Infections and infestations) | 0 | 1 — Not related
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Not related
Blepharospasm (Eye disorders) | 0 | 1 — Not related

LIMITATIONS AND CAVEATS:
This was a pilot study with a small number of subjects not adequately powered to detect treatment differences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Alcon reserves the right of prior review of any publication or presentation of information related to the study.